CLINICAL TRIAL: NCT03620422
Title: Mannitol-Induced Cough Challenge in Healthy Controls and Subjects With Mild Allergic Asthma
Acronym: MICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Syntara (Industry); AllerGen NCE Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: McMaster-MICC4657
Record Dates: First submitted 2018-07-09; First posted 2018-08-08 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2019-03

CONDITIONS: Asthma; Cough
Keywords: Mannitol; Bronchoconstriction; Airway nerve function; Cough; Diagnostic Test; Osmolarity; Salbutamol
MeSH Terms: conditions — Asthma; Cough | interventions — Mannitol; Albuterol; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a mechanistic study. The first part of the study (mild allergic asthmatics and healthy controls) is to determine reproducibility of dose responses to mannitol-induced coughs. The second part of the study (mild asthmatics only) is to determine the effect of salbutamol on mannitol-induced coughs. Salbutamol or placebo will be delivered following a mannitol cough challenge in a randomized, double-blind crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Controls (Other): Mannitol-Induced Cough Challenges on Visit 2 and 3. Mannitol delivered via inhalation. Dosage: 0, 5, 10, 20, 40 mg capsules. 80 and 160 mg doses delivered with two and four capsules, respectively.
  Interventions: Other: Mannitol
- Mild Allergic Asthmatics (Saline) (Placebo Comparator): Mannitol-Induced Cough Challenges on Visit 2, 3 and 4. Nebulized placebo (Sodium Chloride 0.9% Inhl 3Ml) given prior to Mannitol-Induced Cough Challenges on Visit 3 or 4. Mannitol delivered via inhalation. Dosage: 0, 5, 10, 20, 40 mg capsules. 80 and 160 mg doses delivered with two and four capsules, respectively.
  Interventions: Other: Mannitol; Other: Sodium Chloride 0.9% Inhl 3Ml
- Mild Allergic Asthmatics (Salbutamol) (Active Comparator): Mannitol-Induced Cough Challenges on Visit 2, 3 and 4. Nebulized salbutamol (5mg/mL) given prior to Mannitol-Induced Cough Challenges on Visit 3 or 4. Mannitol delivered via inhalation. Dosage: 0, 5, 10, 20, 40 mg capsules. 80 and 160 mg doses delivered with two and four capsules, respectively.
  Interventions: Other: Mannitol; Drug: Salbutamol 5mg/mL

INTERVENTIONS:
Other: Mannitol — Mannitol-Induced Cough Challenge
  Other Names: Aridol
Drug: Salbutamol 5mg/mL — Nebulized salbutamol given prior to Mannitol-Induced Cough Challenge
  Other Names: Active Comparator
  Arms: Mild Allergic Asthmatics (Salbutamol)
Other: Sodium Chloride 0.9% Inhl 3Ml — Nebulized 0.9% saline given prior to Mannitol-Induced Cough Challenge
  Other Names: Placebo Comparator
  Arms: Mild Allergic Asthmatics (Saline)

SUMMARY:
The study aim is to investigate if changes in osmolarity using mannitol challenge can evoke coughing reproducibly in mild allergic asthmatics compared with healthy controls and if salbutamol can affect this. Phase 1 of this study is a reproducibility analysis of cough dose response to mannitol in a cohort of mild allergic asthmatics and healthy controls. Phase 2 is a double-blind, placebo-controlled analysis in mild allergic asthmatics assessing the effects of salbutamol on mannitol induced cough.

DETAILED DESCRIPTION:
The study will have a maximum of 4 visits separated by at least 24 hours. The first 2 visits will determine eligibility. All eligible subjects will be invited back for a third visit, and only subjects with mild allergic asthma will be invited back for a fourth visit.

Screening Period (Visits 1 and 2) - For All Subjects Eligible subjects will be identified during the initial screening procedures with measures of spirometry, hyperresponsiveness to methacholine, complete history, physical examination, allergen skin test, and mannitol cough challenge. The screening procedures will be conducted over 2 separate visits.

Reproducibility (Visit 3) - For Healthy Controls Ten normal healthy controls meeting study eligibility will return for visit 3. This visit must be at least 24h after the mannitol test at visit 1. These data will be used for assessing reproducibility of the mannitol induced coughs; Emax and the median effective dose (ED50).

Effects of Salbutamol (Visit 3 and 4) - For Mild Allergic Asthma Subjects Ten subjects with mild allergic asthma will return for visit 3 and 4. These visits must be at least 24h apart and no longer than 7 days. Mild allergic asthmatics will first receive salbutamol 2.5mg or saline placebo via a nebuliser and 15 mins later the forced expiratory volume at one second (FEV1) measured. Subjects will then undergo a mannitol cough challenge exactly like the previous mannitol cough challenges. These data will be used for determining the effects of salbutamol on mannitol-induced bronchoconstriction and cough.

Visit Windows Each visit must be separated by a minimum of 24 hours, and a maximum of 7 days. Study visits can be performed in the morning or afternoon, however for each subject the timing should be consistent with Visits 2 at the same time of day ± 2 hours

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and give written informed consent
2. Male and female volunteers 18 through 65 years of age.
3. Positive skin-prick test to common aeroallergens (mild allergic asthmatic subjects)
4. Asthma as determined by methacholine provocative concentration causing a 20% fall (PC20) ≤16 mg/ml for mild allergic asthmatic subjects; no airway hyperresponsiveness as determined by methacholine PC20>16mg/ml for normal healthy controls.
5. Baseline FEV1 ≥ 70% of the predicted value for mild allergic asthmatic subjects; baseline FEV1≥ 80% of the predicted value for normal healthy controls.
6. Demonstrate cough response to inhaled mannitol

Exclusion Criteria:

1. Current or former smoker with >10-pack-year history
2. Current or previous history of other significant respiratory disease
3. Significant systemic disease, including history of current malignancy or autoimmune disease
4. Asthma exacerbation or upper/lower respiratory tract infection within the previous 8 weeks
5. Pregnancy
6. Use of corticosteroids within 28 days prior to the first study visit.
7. Use of nonsteroidal anti-inflammatory drugs (NSAIDs) within 48 hours of study visits or aspirin with 7 days of study visits
8. Use of antihistamines including those in cold and allergy medications within 72 hours of study visits
9. Chronic use of other medication for treatment of allergic lung disease other than short-acting β2-agonists.
10. Use of caffeine-containing products within 4 hours of study visits
11. Use of Angiotensin converting enzyme inhibitors (ACE inhibitors)
12. Any centrally acting medication which in the view of the investigator could alter the sensitivity of the cough reflex including but not restricted to tricyclic anti-depressants, pregabalin, gabapentin, codeine, tramadol, or any other opioid.
13. Lung disease other than mild to moderate allergic asthma, for mild allergic asthmatic subjects; no lung disease for normal healthy controls.
14. Unwillingness or inability to comply with the study protocol for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
ED50 dose response curve | Through study completion, an average of one year
  Median effective dose

SECONDARY OUTCOMES:
ED50 (post-bronchodilator) dose response curve | Through study completion, an average of one year
  Median effective dose

CONTACTS AND LOCATIONS:
Overall Officials: Gail Gauvreau, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No